CLINICAL TRIAL: NCT00222729
Title: Phase II Trial of Pemetrexed and Bevacizumab in Patients With Recurrent or Metastatic Head and Neck Cancer
Brief Title: Study of Pemetrexed and Bevacizumab in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-002; 12,158
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: head; neck
MeSH Terms: conditions — Neoplasms | interventions — Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed & Bevacizumab (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 day 1 q 21 days
  Other Names: (N-[4-[2-(2-amino-3,4-dihydron-4-oxo-7H-pyrolo[2,3-d]pyrinidin-5-yl)ethyl]benzoyl]-L-glutamic acid), Alimta, pemetrexed disodium, LY231514, MTA
Drug: Bevacizumab — 15 mg/kg IV q 21 days following pemetrexed
  Other Names: NSC 704865, RhuMAb VEGF, Bevacizumab, Avastin

SUMMARY:
The purpose of this study is to determine if the combination of two new drugs pemetrexed (Alimta) and bevacizumab (Avastin) can increase the effectiveness of treatment for head and neck cancer. Currently pemetrexed is approved by the Food and Drug Administration (FDA) for another type of cancer, mesothelioma, but it is not approved for head and neck cancer.

DETAILED DESCRIPTION:
Main objectives of this study are to 1) evaluate the time to progression (primary endpoint) with the combination of pemetrexed and bevacizumab in recurrent or metastatic head and neck cancer; 2) evaluate the objective response rate, duration of response, overall survival, and toxicities associated with the above therapy and 3) collect tumor tissue from previous diagnostic procedures and blood specimens prospectively, before and after therapy, for future correlative studies.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or locally recurrent squamous cell carcinoma of the head and neck. Patients with local recurrence will be considered incurable by means of locoregional therapy, as judged by the investigator.
2. Cytologically or histologically confirmed squamous cell carcinoma. Nasopharyngeal carcinoma of histologic subtype WHO II and III will be excluded.
3. Unidimensional measurable disease (RECIST criteria). If the only site of measurable disease is in a previously irradiated area, the patient must have documented progression of disease in this area.
4. ECOG performance status 0-1.
5. Full recovered from the effects of any prior surgery, or radiation therapy. A minimum time period of 3 weeks will elapse between the completion of extensive radiation therapy for recurrent/metastatic disease and enrollment in the study
6. Laboratory values:

   ANC ³ 1500/mm³. Platelets ³ 100,000/mm³. Total Bilirubin within normal institutional limits.
7. Transaminases (AST and ALT) < 3 x ULN. Creatinine clearance 45 ml/min or higher calculated using the Cockcroft-Gault formula.
8. Urine protein to creatinine (UPC) ratio of ≤ 1.0 on spot urine urinalysis.
9. Age > 18 years and capacity to give informed consent.

Exclusion Criteria:

1. Prior chemotherapy or biologic therapy for recurrent/metastatic head and neck cancer.
2. Prior pemetrexed, bevacizumab, or other antiangiogenesis agents at any time.
3. Presence of tumors that invaded major vessels.
4. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or anticipation of need for major surgical procedure during the course of the study
5. Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to study enrollment.
6. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration. Serious non-healing wound, ulcer, or bone fracture.
7. History of brain metastasis or seizures.
8. Prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, unless there is a 5-year disease-free interval.
9. Pre-existing peripheral neuropathy > grade 2.
10. Myocardial infarction or stroke in the last 6 months. Unstable angina; Heart Association (NYHA) Grade II or greater congestive heart failure; Clinically significant peripheral vascular disease; CNS cerebrovascular ischemia within the last 6 months; active serious infection; other coexisting medical condition that would preclude full compliance with the study
11. Bleeding diathesis or coagulopathy.
12. Therapeutic anticoagulation (prophylactic use of warfarin 1 mg per day is allowed) or INR greater than 1.5 at registration
13. History of gross hemoptysis (defined as bright red blood of a ½ teaspoon or more).
14. Uncontrolled hypertension (>150/100)
15. Pregnant or lactating.
16. Use of NSAIDs within 5 days of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bauman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Bevacizumab: Patients with previously untreated, recurrent, or metastatic SCCHN treated with pemetrexed 500 mg/m2 and bevacizumab 15 mg/kg
Period: Overall Study
Arm/Group | Pemetrexed + Bevacizumab
Started | 40
Completed | 37
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Bevacizumab
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Time-to-progression (TTP)
Description: TTP was calculated from treatment initiation to disease progression or last follow-up.
Time Frame: Up to 36 months
Population: Evaluable patients with previously untreated, recurrent, or metastatic SCCHN were treated with pemetrexed 500 mg/m2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Bevacizumab
Number analyzed (Participants) | 37
months | 5 [4 to 7]

2. Secondary Outcome: Objective Response Rate (ORR)
Time Frame: Up to 36 months
Population: Evaluable patients with previously untreated, recurrent, or metastatic SCCHN were treated with pemetrexed 500 mg/m2
Measure: Median (90% Confidence Interval); unit: percentage
Arm/Group | Pemetrexed + Bevacizumab
Number analyzed (Participants) | 37
percentage | 30 [17 to 42]

3. Secondary Outcome: Disease Control Rate (DCR)
Time Frame: Up to 36 months
Population: Evaluable patients with previously untreated, recurrent, or metastatic SCCHN were treated with pemetrexed 500 mg/m2 and bevacizumab 15 mg/kg
Measure: Median (90% Confidence Interval); unit: percentage
Arm/Group | Pemetrexed + Bevacizumab
Number analyzed (Participants) | 37
percentage | 86 [77 to 96]

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 36 months
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Bevacizumab
Number analyzed (Participants) | 37
months | 11.3 [8.7 to 16.8]

ADVERSE EVENTS:
Groups:
- Pemetrexed + Bevacizumab: Patients with previously untreated, recurrent, or metastatic SCCHN were treated with pemetrexed 500 mg/m2 and bevacizumab 15 mg/kg
Arm/Group | Pemetrexed + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 28/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed + Bevacizumab (N=40)
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
AST increase (Metabolism and nutrition disorders) | 1
Bleeding (Blood and lymphatic system disorders) | 6
Edema (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 2
Hypertension (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Infection-other (Infections and infestations) | 5
Mucositis (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed + Bevacizumab (N=40)
Constitutional Symptoms - Other (General disorders) | 2
Constitutional Symptoms-Other (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 10
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1
Dysphagia-pharyngeal related to radiation (Gastrointestinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9
Fatigue (asthenia, lethargy, malaise) (General disorders) | 20
Fatigue (lethargy, malaise, asthenia) (General disorders) | 3
Fistula, GI, Oral cavity (Gastrointestinal disorders) | 1
Fistula, GI, Oral cavity (Infections and infestations) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13
Hemoglobin (Blood and lymphatic system disorders) | 13
Hemorrhage, GI, Oral cavity (Blood and lymphatic system disorders) | 2
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 3
Hemorrhage-Other (Blood and lymphatic system disorders) | 1
Hypertension (Vascular disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Infection - Other (Infections and infestations) | 6
Infection without neutropenia (Infections and infestations) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 10
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 4
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Neuropathy: motor (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5
Obstruction/stenosis of airway, Trachea (Respiratory, thoracic and mediastinal disorders) | 1
Pain, Head/headache (General disorders) | 5
Pain-Other (General disorders) | 3
Perforation, GI, Colon (Gastrointestinal disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 2
Seizure (Nervous system disorders) | 1
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 10
Stricture/stenosis (including anastomotic), GI, Esophagus (Gastrointestinal disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Vasovagal episode (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight loss (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No